CLINICAL TRIAL: NCT05942560
Title: Effects of Cognitive Behavioral Therapy-Based Intervention on Depression, Anxiety, Quality of Life, Immune Indicators, and Survival Among Patients With Liver Cancer
Brief Title: Effects of CBT-Based Intervention Among Patients With Liver Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Nethersole School of Nursing (Other)
Collaborators: ZhuHai Hospital (Other)
Responsible Party: Principal Investigator, Hua Yin, Principal Investigator, The Nethersole School of Nursing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CREC2022.328
Record Dates: First submitted 2023-06-25; First posted 2023-07-12 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Depression; Anxiety; Liver Cancer; CBT
Keywords: cognitive behavioural therapy; depression; anxiety; immune; quality of life; survival; liver cancer
MeSH Terms: conditions — Depression; Anxiety Disorders; Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: The study will be a parallel, multicenter, randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: We will ensure that the assessors are unaware of the treatment assignments or intervention details for each participant. We will use anonymized coded data that does not reveal the group allocation during the outcome assessment. The data will be presented in a standardized format that prevents any identification of treatment groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioural therapy-based(CBT-based) intervention group (Experimental): A specifically designed CBT-based intervention consisting of 8 weekly sessions will be conducted in a group format.
  Interventions: Behavioral: Cognitive behavioural therapy-based intervention
- Control group (Active Comparator): Participants will receive eight health education sessions simultaneously with the CBT-based intervention group.
  Interventions: Behavioral: Educational group

INTERVENTIONS:
Behavioral: Cognitive behavioural therapy-based intervention — A specifically designed CBT-based intervention consisting of 8 weekly sessions with group format.
  Each group will be comprised of 4-10 participants, and each session will last 1.5 hours.
  The content of the weekly sessions will be based on Beck's cognitive theory and the cognitive therapy in groups guidelines.
  The framework of every session will follow a pre-determined structure.
  Arms: Cognitive behavioural therapy-based(CBT-based) intervention group
Behavioral: Educational group — The educational sessions are consisting of 8 weekly sessions with a group format. These sessions will focus on cancer-related information and care knowledge which will be delivered in daily routine care.
  Arms: Control group

SUMMARY:
This study investigates the effects of a CBT- based intervention on depression, anxiety, immune function, quality of life, and overall survival. It also explores if the effects of the intervention on immune function and quality of life are mediated through the improvements in depression and anxiety among patients with liver cancer.

DETAILED DESCRIPTION:
In the present research project, the investigators have developed a Cognitive Behavioral Therapy (CBT)-based intervention protocol to investigate the impact of this intervention on depression, anxiety, quality of life, immune function, and overall survival in patients diagnosed with liver cancer. Additionally, this research protocol aims to examine the hypothesized mechanisms underlying the effects of the CBT-based intervention on quality of life and immune function. Specifically, we will investigate: 1) whether the effect of the CBT-based intervention on quality of life is mediated by improvements in anxiety and depression, and 2) whether the effect of the CBT-based intervention on immune function is mediated by improvements in anxiety and depression among patients with liver cancer.

A total of 160 participants will be recruited and randomly assigned to either the CBT-based intervention group or an educational group receiving non-psychological interventions. Assessments will be conducted at baseline (pre-treatment) and at 3, 6, and 12 months after the intervention period. Survival data will be collected throughout the follow-up period until the patients' end-of-life.

By examining the effects of the CBT-based intervention on multiple outcomes and exploring the potential mediating mechanisms, this research project aims to contribute to a comprehensive understanding of the intervention's effectiveness and its impact on the well-being of liver cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (aged ≥18);
2. Diagnosed with liver cancer based on pathological findings or imaging findings in the medical record;
3. The severity level of depression and anxiety: Depression > 7 using HAD-D, or Anxiety > 7 using HAD-A (Hospital Anxiety and Depression Scale, HADS; HAD-D, Hospital Depression Scale; HAD-A, Hospital Anxiety Scale).

Exclusion Criteria:

1. Patients who are taking part in another psychological intervention clinical trial or consented to receive another psychotherapy, suffered from aphasia and other communication difficulties will be excluded from the study
2. Patients with active immunological diseases, such as autoimmune diseases, and inflammatory diseases.
3. Patients accepting hormone therapy or taking long-term antibiotic drugs.
4. Patients who lack the basic ability of understanding and expression and are incompetent in giving consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-12-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Depression symptoms at baseline | T0(Baseline)
  Participants' depression score with the depression subscale of the Hospital depression and Depression Scale (HADS). The HADS depression subscale score ranges from 0 to 21, with higher scores indicating more severe depression symptoms.
Change in depression symptoms at 3 months | T1(3 months)
  Change in participants' depression score with the HADS depression subscale from baseline to 3 months. The HADS depression subscale score ranges from 0 to 21, with higher scores indicating more severe depression symptoms.
Change in depression symptoms at 6 months | T2(6 months)
  Change in participants' depression score with the HADS depression subscale from baseline to 6 months. The HADS depression subscale score ranges from 0 to 21, with higher scores indicating more severe depression symptoms.
Change in depression symptoms at 12 months | T3(12 months)
  Change in participants' depression score with the HADS depression subscale from baseline to 12 months. The HADS depression subscale score ranges from 0 to 21, with higher scores indicating more severe depression symptoms.
Anxiety symptoms at baseline | T0(Baseline)
  Participants' anxiety score with the Anxiety subscale of the Hospital Anxiety and Depression Scale (HADS). The HADS anxiety subscale score ranges from 0 to 21, with higher scores indicating more severe anxiety symptoms.
Change in anxiety symptoms at 3 months | T1(3 months)
  Change in participants' anxiety score with the HADS anxiety subscale from baseline to 3 months. The HADS anxiety subscale score ranges from 0 to 21, with higher scores indicating more severe anxiety symptoms.
Change in anxiety symptoms at 6 months | T2(6 months)
  Change in participants' anxiety score with the HADS anxiety subscale from baseline to 6 months. The HADS anxiety subscale score ranges from 0 to 21, with higher scores indicating more severe anxiety symptoms.
Change in anxiety symptoms at 12 months | T3(12 months)
  Change in participants' anxiety score with the HADS anxiety subscale from baseline to 12 months. The HADS anxiety subscale score ranges from 0 to 21, with higher scores indicating more severe anxiety symptoms.

SECONDARY OUTCOMES:
Quality of life score (The EORTC QLQ-C30) at baseline | T0(Baseline)
  The European Organization for Research and Treatment of Cancer(EORTC) Quality of Life Questionnaire results.
  Scores range from 0 to 100. A higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
Change in Quality of life score (The EORTC QLQ-C30) at 3 months | T1(3 months)
  The European Organization for Research and Treatment of Cancer(EORTC) Quality of Life Questionnaire results.
  Scores range from 0 to 100. A higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
Change in Quality of life score (The EORTC QLQ-C30) at 6 months | T2(6 months)
  The European Organization for Research and Treatment of Cancer(EORTC) Quality of Life Questionnaire results.
  Scores range from 0 to 100. A higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
Change in Quality of life score (The EORTC QLQ-C30) at 12 months | T3(12 months)
  The European Organization for Research and Treatment of Cancer(EORTC) Quality of Life Questionnaire results.
  Scores range from 0 to 100. A higher score represents a higher ("better") level of functioning, or a higher ("worse") level of symptoms.
Quality of life score (The EORTC QLQ-HCC18) at baseline | T0(Baseline)
  The Hepatocellular Carcinoma Module of The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire. Scores range from 0 to 100. A higher score represents a high level of symptomatology or problems.
Change in Quality of life score (The EORTC QLQ-HCC18) at 3 months | T1(3 months)
  The Hepatocellular Carcinoma Module of The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire. Scores range from 0 to 100. A higher score represents a high level of symptomatology or problems.
Change in Quality of life score (The EORTC QLQ-HCC18) at 6 months | T2(6 months)
  The Hepatocellular Carcinoma Module of The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire. Scores range from 0 to 100. A higher score represents a high level of symptomatology or problems.
Change in Quality of life score (The EORTC QLQ-HCC18) at 12 months | T3(12 months)
  The Hepatocellular Carcinoma Module of The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire. Scores range from 0 to 100. A higher score represents a high level of symptomatology or problems.
Immune variables 1 at baseline | T0(Baseline)
  Total lymphocyte count. Collected from daily medical records.
Change in Immune variables 1 at 3 months | T1(3 months)
  Total lymphocyte count. Collected from daily medical records.
Change in Immune variables 1 at 6 months | T2(6 months)
  Total lymphocyte count. Collected from daily medical records.
Immune variables 2 at baseline | T0(Baseline)
  Level of IFN-γ. Collected from blood sample.
Change in Immune variables 2 at 3 months | T1(3 months)
  Level of IFN-γ. Collected from blood sample.
Change in Immune variables 2 at 6 months | T2(6 months)
  Level of IFN-γ. Collected from blood sample.
Immune variables 3 at baseline | T0(Baseline)
  IL-2. Collected from blood sample.
Change in Immune variables 3 at 3 months | T1(3 months)
  IL-2. Collected from blood sample.
Change in Immune variables 3 at 6 months | T2(6 months)
  IL-2. Collected from blood sample.
Immune variables 4 at baseline | T0(Baseline)
  IL-4. Collected from blood sample.
Change in Immune variables 4 at 3 months | T1(3 months)
  IL-4. Collected from blood sample.
Change in Immune variables 4 at 6 months | T2(6 months)
  IL-4. Collected from blood sample.
Immune variables 5 at baseline | T0(Baseline)
  IL-6. Collected from blood sample.
Change in Immune variables 5 at 3 months | T1(3 months)
  IL-6. Collected from blood sample.
Change in Immune variables 5 at 6 months | T2(6 months)
  IL-6. Collected from blood sample.
Overall survival | T3 (12 months) and later till the end of life.
  Survival status form follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Hua Yin, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Zhuhai People's Hospital, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No